CLINICAL TRIAL: NCT06406595
Title: Hemispheric Asymmetries in Emotion-Cognition Interactions
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00130303
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Anxiety Depression Disorder
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older Adults Healthy Control Group: The healthy older adult group is carefully defined to serve as a comparison group against individuals with mental health issues. By selecting participants aged over 60 who do not exhibit mental health issues and demonstrate healthy aging from a cognitive perspective, the investigators establish a baseline for cognitive functioning within the older adult population.
  Interventions: Other: Observation
- Older Adults with Mental Health Issues Group: The older adults with mental health issues group is crucial for examining the impact of Anxiety and/or Depression on cognitive aging. Participants aged over 60 diagnosed with these conditions are included while still demonstrating healthy aging from a cognitive standpoint. This ensures that any observed cognitive differences can be attributed to mental health conditions rather than age-related decline alone.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — This study is observational, therefore, there is no intervention included.

SUMMARY:
In this research, the investigators will recruit 2 groups of individuals: older adults (aged over 65) with anxiety and/or depression and older adults without mental health issues. Individuals who are eligible to participate in the study based on their score in the Edinburgh Handedness Inventory (EHI) showing their hand preferences will have the opportunity to sign up using the online form created by the research team. This experiment will take place in an electroencephalogram (EEG) lab. Participants will wear an EEG cap with 256 sensors that record their brain activity while completing an emotional oddball task containing emotional pictures and shapes. The task will take approximately 1 hour with 8 short breaks. EEG is a safe and non-invasive testing technique, and participants will feel little or no discomfort during this EEG experiment. The goal of this study is to investigate the effect of fearful emotion on the cognitive oddball task to deepen understanding of the emotion-cognition interaction in older adults with mental health conditions.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of fearful emotion on the cognitive oddball task using electroencephalogram (EEG) technology. The study aims to deepen the understanding of the emotion-cognition interaction in humans. Emotions are fundamental to human behavior, and they can have a significant impact on cognitive processes such as attention, memory, and decision-making. Furthermore, the relationship between emotion and cognition has been implicated in numerous psychiatric disorders, including anxiety, depression, and post-traumatic stress disorder. Therefore, understanding the mechanisms by which emotions affect cognition is essential for the development of effective treatments for these disorders.

Electroencephalography (EEG) is a non-invasive and widely-used technique that measures the electrical activity of the brain, making it an excellent tool for studying the relationship between emotion and cognition. This study will use EEG to examine the neural correlates of attentional processing in response to emotional stimuli. Specifically, the investigators will use an emotional oddball task to investigate the effect of fearful emotions on the attention of deviant stimuli, which is an established paradigm in the study of emotion and cognition.

Furthermore, this study will explore the impact of the location of the deviant stimuli presentation (i.e., in the left or right visual field) on the emotion-cognition interaction. This variable is crucial because previous research has suggested hemispheric asymmetries in emotion processing and contralateral visual processing. By including this variable in the study, the investigators will be able to examine whether the emotion-cognition interaction is influenced by the location of stimulus presentation.

Additionally, the investigators will include 2 groups: older adults with anxiety and/or depression, and older adults without mental health issues. By examining these different groups, the investigators aim to elucidate how mental health status may modulate emotion-cognition interactions.

The inclusion of novel variables, such as the location of stimulus presentation and mental health status, makes this study innovative and likely to produce novel findings that will contribute to the existing literature on this topic. It is hypothesized that the presentation of fearful images in the cognitive oddball task will result in greater changes in brain electrical activity as compared to neutral images. Specifically, the investigators expect to observe increased activity in the ventral affective system (e.g., amygdala) and other regions of the brain associated with emotional processing. The investigators also hypothesize that the location of the shape presentation (whether on the left or right visual field) may modulate the effect of emotion on cognition by influencing the event-related potentials (ERPs) in dorsal executive system (e.g., dorsal lateral prefrontal cortex (dlPFC)).

The objectives of this study are:

* To investigate the effect of fearful emotion on the cognitive oddball task using EEG technology.
* To analyze changes in brain electrical activity in response to fearful and neutral stimuli.
* To investigate whether the location of shape presentation (left or right visual field) modulates the effect of emotion on cognition.
* To explore how mental health status may modulate emotion-cognition interactions.

Research Method/Procedures:

Participants who meet the inclusion criteria (strong handedness) will be scheduled for a one-hour session in the EEG lab. During the session, participants will wear an EEG cap with 256 channels that record their brain electrical activity while they complete an emotional oddball task. The task will consist of fearful and neutral pictures and black circles that are shown in the middle, left, or right visual field of the screen. The frequency of shapes appearing in the left or right visual field will be varied to investigate the impact of visual field location. The task duration will be approximately 1 hour with 8 short breaks during the processing.

For data analysis, the investigators will analyze the EEG data using time-frequency analysis to identify changes in brain electrical activity in response to fearful and neutral stimuli. The investigators will compare the results of the odd stimulus after fearful images with that after neutral images to isolate the effect of emotions on cognitive processing. The investigators will also use statistical analysis to identify any significant differences in the impact of visual field location on the effect of emotion on cognition. Finally, the investigators will interpret our findings in the context of existing literature on the emotion-cognition interaction in humans, and conduct cross-sectional comparisons between different mental health conditions to investigate the generalizability of the findings.

ELIGIBILITY:
Inclusion Criteria:

* The healthy older adult group is composed of participants aged over 60 who do not exhibit mental health issues and demonstrate healthy aging from a cognitive perspective.
* The older adults with mental health issues group will consist participants aged over 60 diagnosed with these conditions are included while still demonstrating healthy aging from a cognitive standpoint.

Exclusion Criteria:

* Participants currently taking medication known to affect brain activity and/or cognitive processing.
* Participants with a history of alcohol or substance abuse.
* Participants with a history of head injury or concussion that may impact brain activity and/or cognitive processing.
* Participants with Neurological Disorders.
* Participants with Edinburgh Handedness Inventory scores falling within the range of [-40, 40].

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Healthy older adult aged over 60 who do not exhibit mental health issues and demonstrate healthy aging from a cognitive perspective.
  2. Older adults aged over 60 who have been diagnosed with Anxiety and/or Depression, while still demonstrating healthy aging from a cognitive standpoint.
  Participants with Edinburgh Handedness Inventory scores falling within the range of [-100, -41] and [41, 100] are eligible to participate in this study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Event-related potentials(ERPs): Peak Amplitude of P100, P300, and Late Positive Potential | After the raw EEG data being collected, the investigators plan to conduct preprocessing, independent component analysis and extract ERPs of our interest starting in January 2025.
  This study investigates Event-Related Potentials (ERPs), focusing on P100, P300, and Late Positive Potential (LPP). The peak amplitude of these components reflects the maximum voltage deflection recorded from the scalp during these time windows following specific stimuli. By analyzing the peak amplitude, the investigators aim to explore the neural mechanisms implicated in cognitive functions such as attention, decision-making, and emotional processing.
Event-related potentials(ERPs): Latency of P100, P300, and Late Positive Potential | After the raw EEG data being collected, the investigators plan to conduct preprocessing, independent component analysis and extract ERPs of our interest starting in January 2025.
  This study investigates Event-Related Potentials (ERPs), focusing on P100, P300, and Late Positive Potential (LPP). The latency of these components represents the time between the presentation of a stimulus and the peak activity they exhibit. The value of latency lies in its precision regarding the timing of cognitive processes. Through latency analysis, the investigators gain a detailed understanding of the sequential progression of neural events.
Magnitude of Rhythmic Activity in EEG Oscillations: Alpha, Theta, and Delta Bands | After the raw EEG data being collected, the investigators plan to conduct preprocessing, independent component analysis and extract EEG bands of our interest starting in January 2025.
  This study explores emotion and visual attention aspects within EEG oscillations, particularly in the Alpha, Theta, and Delta bands. These bands are known to influence emotional processing and attentional mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Singhal, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada